CLINICAL TRIAL: NCT02864576
Title: Cognitive Remediation Plus Aerobic Exercise in Schizophrenia Treatment: a Randomized Controlled Study.
Brief Title: Cognitive Remediation Plus Aerobic Exercise in Schizophrenia Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Nuria Pujol, Clinical Psychologist, Principal Investigator, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI15/00453
Record Dates: First submitted 2016-07-26; First posted 2016-08-12 (Estimated); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Remediation_Aerobic Exercise (Experimental): Cognitive Remediation:
  12 weeks of systematic cognitive training (REHACOP), performed 3 days per week in a 90-minutes-long sessions.
  Aerobic Exercise:
  12 weeks of systematic aerobic exercise program, performed 3 days per week, lasting 40 minutes.
  Interventions: Behavioral: Cognitive Remediation_Aerobic Exercise
- Cognitive Remediation_Health Promotion (Active Comparator): Cognitive Remediation:
  12 weeks of systematic cognitive training (REHACOP), performed 3 days per week in a 90-minutes-long sessions.
  Health Promotion:
  12 weeks of health promotion sessions, performed 3 days per week, lasting 40 minutes each.
  Interventions: Behavioral: Cognitive Remediation_Health Promotion

INTERVENTIONS:
Behavioral: Cognitive Remediation_Aerobic Exercise — Cognitive Remediation:
  The REHACOP program consists of: Attention unit training sustained, selective, alternant and divided attention; Memory unit focusing on visual and verbal learning, recall and recognizing memory; Language unit including grammar, syntax, vocabulary, verbal fluency, verbal comprehension, abstract language; Executive functions unit training cognitive planning, proverbs, analogies; and Social cognition unit exercising theory of mind, social reasoning and moral dilemmas.
  Aerobic Exercise:
  12 weeks of systematic aerobic exercise program. Patients will walk with a moderate intensity 10 minutes the first week and will increase gradually up to 30 minutes-walk with a moderate intensity. Patients will also perform 5 minutes of warm-up and stretching.
  Arms: Cognitive Remediation_Aerobic Exercise
Behavioral: Cognitive Remediation_Health Promotion — Cognitive Remediation:
  The REHACOP program consists of: Attention unit training sustained, selective, alternant and divided attention; Memory unit focusing on visual and verbal learning, recall and recognizing memory; Language unit including grammar, syntax, vocabulary, verbal fluency, verbal comprehension, abstract language; Executive functions unit training cognitive planning, proverbs, analogies; and Social cognition unit exercising theory of mind, social reasoning and moral dilemmas.
  Health Promotion:
  12 weeks of health promotion sessions. These sessions will be carried out by a specialized/trained nurse.
  Other Names: Cognitive Remediation_Control Activity
  Arms: Cognitive Remediation_Health Promotion

SUMMARY:
Cognitive remediation (CR) and aerobic exercise have separately shown promising results in schizophrenia cognitive improvement, despite this, the impact in improving functionality is still limited. Aerobic exercise increases Brain Derived Neurotrophic Factor (BDNF) levels, promoting neuronal and cognitive plasticity, which can maximize the impacts of CR. The aim of this randomized controlled trial is to study the efficacy of a 3-month intensive program that combines CR plus physical exercise comparing it to cognitive remediation plus a control activity.

DETAILED DESCRIPTION:
Cognitive remediation (CR) and physical exercise have separately shown promising results in schizophrenia cognitive improvement, despite this, the impact in improving functionality is still limited. Physical exercise increases Brain Derived Neurotrophic Factor (BDNF) levels, promoting neuronal and cognitive plasticity, which can maximize the impact of CR. The aim of this project is to study the efficacy of an intensive program (3 months) that combines CR and physical exercise by a randomized controlled trial where 74 patients with chronic schizophrenia will be randomized to two groups: 1) CR plus physical exercise; 2) CR plus control activity (health promotion). Primary outcome measures will be cognitive performance, functional outcome, negative symptoms and BDNF levels. Measures will be blindly assessed at baseline, at 3 months follow up and at 15 months follow up. The investigators expect that: i) the CR plus physical exercise will be superior to CR plus control activity in improving cognition, functional outcome, negative symptoms and in increasing BDNF levels in the short and medium term (3 and 15 months); ii) changes in BDNF levels after the CR plus physical exercise will be an adequate biomarker of the cognitive improvement obtained with this treatment.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis by Diagnostic and Statistical Manual of Mental Disorders of schizophrenia or schizoaffective disorder with a minimum of 10 years illness evolution/duration;
2. Between 28 and 60 years of age;
3. Clinically stable (no changes in psychotropic medication in the previous months, except for benzodiazepines)
4. Sufficient acculturation and fluency in the Spanish language to avoid invalidating research measures of thought, language, and speech disorder or of verbal cognitive abilities;
5. Low physical activity, as measured by International Physical Activity Questionnaire, IPAQ;
6. Signed informed consent

Exclusion Criteria:

1. Evidence of a known neurological disorder (e.g., epilepsy) or significant head injury;
2. Evidence of substance use disorder within the previous 3 months;
3. mental retardation, i.e. premorbid intelligence quotient less than 70;
4. Electroconvulsive therapy in previous 6 months.
5. Somatic illnesses that contraindicate physical exercise.

Ages: 28 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2016-09; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) overall composite score | 3 months

SECONDARY OUTCOMES:
Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) overall composite score | 15 months
Brain-derived neurotrophic factor (BDNF) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Núria Pujol, PhD, Principal Investigator — Parc de Salut Mar, Barcelona, Spain; Anna Mané, MD, PhD, Principal Investigator — Parc de Salut Mar, Barcelona, Spain
Locations (1):
- Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No